CLINICAL TRIAL: NCT06317662
Title: A Phase 2 Study of Blinatumomab in Combination With Chemotherapy for Infants With Newly Diagnosed Acute Lymphoblastic Leukemia With Randomization of KMT2A-Rearranged Patients to Addition of Venetoclax
Brief Title: Testing the Addition of the Anti-cancer Drug Venetoclax and/or the Anti-cancer Immunotherapy Blinatumomab to the Usual Chemotherapy Treatment for Infants With Newly Diagnosed KMT2A-rearranged or KMT2A-non-rearranged Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01994; NCI-2024-01994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL2321 (Other: Children's Oncology Group); AALL2321 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2024-03-16; First posted 2024-03-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia of Ambiguous Lineage; B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Burkitt Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; calaspargase pegol; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Levoleucovorin; Spinal Puncture; Magnetic Resonance Spectroscopy; Mercaptopurine; azathiopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; Prednisolone; Prednisone; deltacortene; prednylidene; Hydrocortisone; Thioguanine; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm A (Experimental): See Detailed Description for Arm A.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine
- Arm B, Cohort 1 (Experimental): See Detailed Description for Arm B, Cohort 1.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine
- Arm B, Cohort 2 (Experimental): See Detailed Description for Arm B, Cohort 2.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine
- Arm B, Cohort 3 (Experimental): See Detailed Description for Arm B, Cohort 3.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine
- Arm B, Cohort 4 (Experimental): See Detailed Description for Arm B, Cohort 4.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine
- Arm C (Experimental): See Detailed Description for Arm C.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Methylprednisolone; Procedure: Multigated Acquisition Scan; Drug: Prednisolone; Drug: Prednisone; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine
- Safety Phase Cohort (Experimental): See Detailed Description for Safety Phase Cohort.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Drug: Leucovorin; Drug: Levoleucovorin; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine
- Steroid Prephase(prednisone, prednisolone, methylprednisolone) (Experimental): All patients receive prednisone or prednisolone PO or NG TID or methylprednisolone IV TID for 7 days prior to the start of induction therapy (on days 1-7).
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: FDG-Positron Emission Tomography; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Methylprednisolone; Procedure: Multigated Acquisition Scan; Drug: Prednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given recombinant crisantaspase IM or crisantaspase IM or IV
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Safety Phase Cohort
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Dexamethasone — Given PO or NG or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Arm C
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Drug: Leucovorin — Given PO or NG or IV
  Other Names: Folinic acid
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Levoleucovorin — Given IV
  Other Names: CL-307,782; Elvorine, Isovorin, Levofolene, Levorin; Isovorin; L-Leucovorin; Levofolinate; Levofolinic acid
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mercaptopurine — Given PO or NG
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Methotrexate — Given IT or IV or PO or NG
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
  Arms: Arm C; Steroid Prephase(prednisone, prednisolone, methylprednisolone)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Prednisolone — Given PO or NG
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: Arm C; Steroid Prephase(prednisone, prednisolone, methylprednisolone)
Drug: Prednisone — Given PO or NG
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm C; Steroid Prephase(prednisone, prednisolone, methylprednisolone)
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Thioguanine — Given PO or NG
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort
Drug: Venetoclax — Given PO or NG
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Safety Phase Cohort
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Arm A; Arm B, Cohort 1; Arm B, Cohort 2; Arm B, Cohort 3; Arm B, Cohort 4; Arm C; Safety Phase Cohort

SUMMARY:
This phase II trial tests the addition of venetoclax and/or blinatumomab to usual chemotherapy for treating infants with newly diagnosed acute lymphoblastic leukemia (ALL) with a KMT2A gene rearrangement (KMT2A-rearranged [R]) or without a KMT2A gene rearrangement (KMT2A-germline [G]). Venetoclax is in a class of medications called B-cell lymphoma-2 (Bcl-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Blinatumomab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding venetoclax and/or blinatumomab to standard chemotherapy may be more effective at treating patients with ALL than standard chemotherapy alone, but it may also cause more side effects. This clinical trial evaluates the safety and effectiveness of adding venetoclax and/or blinatumomab to chemotherapy for the treatment of infants with KMT2A-R or KMT2A-G ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of venetoclax in addition to a standard chemotherapy backbone and two cycles of blinatumomab in infants (aged 365 days or less at diagnosis) with newly diagnosed KMT2A-R ALL.

II. To determine in a randomized manner if the addition of venetoclax to induction chemotherapy improves end of induction minimal residual disease (MRD)-negative remission rates in infants with KMT2A-R ALL.

SECONDARY OBJECTIVES:

I. To estimate the MRD-negative remission rate for all eligible infants with KMT2A-R ALL treated with venetoclax at the recommended phase 2 dose (RP2D).

II. To compare event free survival (EFS) rates of infants with KMT2A-R ALL treated on arm B to those treated on arm A.

III. To compare 3-year EFS rates of infants with KMT2A-R ALL treated on arm A to historical controls.

IV. To determine the feasibility of treating infants with KMT2A-G ALL with a Children's Oncology Group (COG) high risk ALL chemotherapy backbone and two cycles of blinatumomab and estimate the 3-year EFS rate of infants with KMT2A-G ALL treated on arm C.

V. To characterize the pharmacokinetics (PK) of venetoclax in infants.

EXPLORATORY OBJECTIVES:

I. To describe 3-year EFS rate of infants with KMT2A-R ALL treated on arm B. II. To evaluate the use of high-throughput sequencing (HTS) for MRD detection in infant ALL compared to centralized flow cytometry.

III. To characterize the PK of calaspargase pegol-mknl in infants with ALL. IV. To report the incidence of CD19 negative relapse and myeloid switch relapse with protocol therapy.

V. To evaluate the impact of venetoclax in combination with chemotherapy on T-cell subsets and function.

VI. To describe the feasibility of T-cell collection and success of T-cell manufacturing for infants with KMT2A-R ALL who receive chimeric antigen receptor (CAR) T- cell therapy after coming off protocol therapy.

VII. To determine predictors of response and resistance to venetoclax and overall protocol therapy.

VIII. To evaluate the impact of subsequent anti-cancer therapy on overall survival after coming off protocol therapy.

OUTLINE:

STEROID PREPHASE: All patients receive prednisone or prednisolone orally (PO) or nasogastrically (NG) three times daily (TID) or methylprednisolone intravenously (IV) TID for 7 days prior to the start of induction therapy (on days 1-7).

Patients who are KMT2A gene rearrangement positive are assigned to the safety phase cohort during the safety phase of the study, or randomized between Arm A and Arm B during the expansion phase of the study. Patients who are KMT2A gene rearrangement negative are assigned to Arm C.

SAFETY PHASE COHORT:

INDUCTION: Patients receive venetoclax PO or NG once daily (QD) on days 1-7, 1-10, or 1-14, daunorubicin IV over 1-15 minutes on days 1 and 2, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy (methotrexate, hydrocortisone, cytarabine) intrathecally (IT) on days 1, 15, and 29 or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when absolute neutrophil counts (ANC) >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-central nervous system (CNS) extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine subcutaneously (SC) QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

EXPANSION PHASE: After completion of Safety phase, patients who are KMT2A gene rearrangement positive are randomized to Arm A or Arm B.

ARM A:

INDUCTION: Patients receive daunorubicin IV over 1-15 minutes on days 1 and 2, cytarabine SC or IV over 15-30 minutes on days 1-14, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29, or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

ARM B: Patients are assigned to 1 of 4 cohorts.

COHORT 1:

INDUCTION + VENETOCLAX: Patients receive venetoclax PO or NG QD, daunorubicin IV over 1-15 minutes on days 1 and 2, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29 or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA + VENETOCLAX: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, venetoclax PO or NG QD, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

COHORT 2:

INDUCTION + VENETOCLAX: Patients receive venetoclax PO or NG QD, daunorubicin IV over 1-15 minutes on days 1 and 2, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29 or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION + VENETOCLAX: Patients receive venetoclax PO or NG QD, cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

COHORT 3:

INDUCTION + VENETOCLAX: Patients receive venetoclax PO or NG QD, daunorubicin IV over 1-15 minutes on days 1 and 2, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29 or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION + VENETOCLAX: Patients receive venetoclax PO or NG QD, cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA + VENETOCLAX: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, venetoclax PO or NG QD, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

COHORT 4:

INDUCTION + VENETOCLAX: Patients receive venetoclax PO or NG QD, daunorubicin IV over 1-15 minutes on days 1 and 2, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29 or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and intrathecal therapy IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, and intrathecal therapy IT on day 29. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to MARMA the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MARMA: Patients receive mercaptopurine PO or NG QD on days 1-14, high dose methotrexate IV over 24 hours on days 1 and 8, leucovorin PO, NG, or IV or levoleucovorin IV on days 3-4 and 10-11, intrathecal therapy IT on days 1 and 8, high dose cytarabine IV over 3 hours on days 22-23 and 29-30, and recombinant crisantaspase IM or crisantaspase IM or IV over 1-2 hours on days 23 and 30. At the end of MARMA (day 49), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28 and intrathecal therapy IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive calaspargase pegol IV over 1-2 hours on day 1, dexamethasone PO, NG, or IV TID on days 1-21, thioguanine PO or NG on days 1-28 and 36-49, vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine SC or IV over 15-30 minutes on days 2-5, 9-12, 16-19, 23-26, 37-40, and 44-47, cyclophosphamide IV over 15-30 minutes on days 36 and 50, and intrathecal therapy IT on days 1 and 15. At the end of delayed intensification (day 63), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

MAINTENANCE: Patients receive mercaptopurine PO or NG on days 1-84 of each cycle, methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and intrathecal therapy IT on day 1 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of MARMA in the absence of disease progression or unacceptable toxicity.

ARM C:

INDUCTION: Patients receive daunorubicin IV over 1-15 minutes on days 1 and 2, cytarabine SC or IV over 15-30 minutes on days 1-14, vincristine IV on days 1, 8, 15, and 22, dexamethasone PO, NG, or IV TID on days 1-28, calaspargase pegol IV over 1-2 hours on day 4, and intrathecal therapy IT on days 1, 15, and 29, or days 1, 8, 15, 22, and 29. Patients with < 5% blasts by morphology in the bone marrow at the end of induction (day 35) proceed directly to blinatumomab block 1 on the next day or when ANC >= 500/uL and platelets >= 50,000/uL. Patients with >= 5% blasts by morphology in the bone marrow at the end of induction proceed to blinatumomab block 1 as soon as marrow results are known, irrespective of ANC or platelet values.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO, NG, or IV on day 1 or days 1 and 8, blinatumomab IV on days 1-28, 1-7, or 8-28, and methotrexate IT on days 15 and 29. Patients who are MRD >= 1% or who have residual non-CNS extramedullary disease at the end of blinatumomab block 1 (day 35) discontinue protocol therapy. All other patients proceed directly to consolidation on the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine SC QD or IV over 15-30 minutes on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO or NG QD on days 1-14 and 29-42, methotrexate IT on days 8, 15, and 22, vincristine IV on days 15, 22, 43, and 50, and calaspargase pegol IV over 1-2 hours on days 15 and 43. Patients who are MRD >= 0.01% at the end of consolidation therapy (day 56) discontinue protocol therapy. All other patients proceed directly to interim maintenance 1 the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

INTERIM MAINTENANCE 1: Patients receive vincristine IV on days 1, 15, 29, and 43, high dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, mercaptopurine PO or NG on days 1-14, 15-28, 29-42, and 43-56, methotrexate IT on days 1 and 29, and leucovorin PO or NG or IV or levoleucovorin IV on days 3-4, 17-18, 31-32, and 45-46. At the end of interim maintenance 1 (day 63), all patients proceed directly to blinatumomab block 2 the next day or when peripheral counts recover to ANC >= 500/uL and platelets >= 50,000/uL.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV on days 1-28, and methotrexate IT on days 1 and 15. At the end of blinatumomab block 2 (day 35), all patients proceed directly to delayed intensification the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

DELAYED INTENSIFICATION: Patients receive methotrexate IT on days 1, 29, and 36, dexamethasone PO, NG, or IV TID on days 1-7 and 15-21, vincristine IV on days 1, 8, 15, 43, and 50, doxorubicin IV over 3-15 minutes on days 1, 8, and 15, calaspargase pegol IV over 1-2 hours on days 4 and 43, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO or NG on days 29-42, and cytarabine SC or IV over 15-30 minutes on days 29-32 and 36-39. At the end of delayed intensification (day 63), all patients proceed directly to interim maintenance 2 the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

INTERIM MAINTENANCE 2: Patients receive vincristine IV on days 1, 11, 21, 31, and 41, methotrexate IV push over 2-5 minutes of IV over 10-15 minutes on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and calaspargase pegol IV over 1-2 hours on days 2 and 23. At the end of interim maintenance 2 (day 56), all patients proceed directly to maintenance the next day or when peripheral counts recover to ANC >= 750/uL and platelets >= 75,000/uL.

MAINTENANCE: Patients receive methotrexate IT on day 1 of each cycle, vincristine IV on day 1 of each cycle, prednisone or prednisolone PO or NG BID or methylprednisolone IV BID on days 1-5 of each cycle, mercaptopurine PO or NG on days 1-84 of each cycle, and methotrexate PO, NG, or IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 of each cycle. Cycles repeat every 12 weeks (84 days) for up to 2 years from the start of interim maintenance 1 in the absence of disease progression or unacceptable toxicity.

All patients undergo bone marrow aspiration, collection of blood samples and echocardiography (ECHO) or multigated acquisition scan (MUGA) throughout the trial. Patients may undergo computed tomography (CT), magnetic resonance imaging (MRI), fludeoxyglucose-positron emission tomography (FDG-PET), and/or lumbar puncture if clinically indicated.

After completion of study treatment, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be enrolled on APEC14B1 and consented to eligibility screening (part A) prior to treatment and enrollment on AALL2321
* Infants (aged 365 days or less) on the date of diagnosis are eligible; infants must be > 36 weeks gestational age at the time of enrollment
* Patients must have newly diagnosed B-acute lymphoblastic leukemia (B-ALL, 2017 World Health Organization [WHO] classification), also termed B-precursor ALL, or acute leukemia of ambiguous lineage (ALAL), which includes mixed phenotype acute leukemia. For patients with ALAL, the immunophenotype of the leukemia must comprise at least 50% B lineage

  * Diagnostic immunophenotype: Leukemia cells must express CD19

Exclusion Criteria:

* Patients with Down Syndrome
* Patients with secondary B-ALL that developed after treatment of a prior malignancy with cytotoxic chemotherapy
* Patients must not have received any cytotoxic chemotherapy for either the current diagnosis of infant ALL or for any cancer diagnosis prior to the initiation of protocol therapy, with the exception of:

  * Steroid pretreatment:

    * PredniSONE, prednisoLONE, or methylPREDNISolone for ≤ 72 hours (3 days) in the 7 days prior to enrollment. The dose of predniSONE, prednisoLONE or methylPREDNISolone does not affect eligibility
    * Inhaled and topical steroids are not considered pretreatment
    * Note: Pretreatment with dexamethasone in the 28 days prior to initiation of protocol therapy is not allowed with the exception of a single dose of dexamethasone used during or within 6 hours prior to or after sedation to prevent or treat airway edema. However, prior exposure to ANY steroids that occurred > 28 days before enrollment does not affect eligibility
  * Intrathecal cytarabine or methotrexate:

    * An intrathecal dose of cytarabine or methotrexate in the 7 days prior to enrollment does not affect eligibility
    * Note: The preference is to defer the diagnostic lumbar puncture with intrathecal chemotherapy to day 1 of induction to allow for cytoreduction of circulating blasts and decrease the potential for central nervous system (CNS) contamination due to a traumatic tap. If done prior to day 1 of induction, these results will be used to determine CNS status
  * Hydroxyurea:

    * Pretreatment with ≤ 72 hours (3 days) of hydroxyurea in the 7 days prior to enrollment does not affect eligibility
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA) and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) (safety phase) | For the duration of the induction + venetoclax cycle
  For the safety phase, DLTs of the induction + venetoclax cycle of KMT2A-rearranged (R) patients will be assessed.
Incidence of DLTs (expansion phase) | During the induction, consolidation, and MARMA cycles of Arm B
  For the expansion phase, DLTs of Arm B will be assessed and monitored for the cycles that contain venetoclax (induction, consolidation, and MARMA cycles of Arm B).
Minimal residual disease (MRD)-negative remission rate | At the end of induction
  The end of induction MRD-negative remission rate will be compared between Arm A and Arm B. MRD negativity is defined as achievement of complete remission and MRD < 0.01% by flow cytometry. The MRD-negative remission rate at the end of induction between Arm A and Arm B will be compared using a one-sided Z test of proportions with Type I error of 0.15.

SECONDARY OUTCOMES:
MRD-negative remission rate | At the end of induction
  MRD-negative remission rate at the end of induction and the standard error or 95% confidence interval will be estimated among infants with KMT2A-R acute lymphoblastic leukemia (ALL) treated with venetoclax at the RP2D. This analysis will include eligible KMT2A-R patients treated with venetoclax at the RP2D in the safety phase, as well as patients randomized to Arm B and treated with venetoclax in the expansion phase. MRD negativity is defined as < 0.01% by flow cytometry.
Event free survival (EFS) rates of infants with KMT2A-R ALL | From date of randomization to treatment failure, first documented relapse following achievement of remission-1, occurrence of a second or secondary malignant neoplasm, or death, assessed up to 3 years
  The EFS rates from date of randomization of Arm B will be compared to Arm A. Comparison of EFS rates between Arm A and Arm B will be based on a one-sided logrank test with Type I error of 0.15.
3-year EFS of infants with KMT2A-R ALL | From date of randomization to treatment failure, first documented relapse following achievement of remission-1, occurrence of a second or secondary malignant neoplasm, or death, assessed up to 3 years
  For Arm A, the 3-year EFS rate (representing a plateau rate based on the shape of EFS curves of historical data in this patient population) from the date of randomization will be compared to the stable historical 3-year EFS rate of 35% observed in AALL0631 and other international trials.
Proportion of KMT2A-germline (G) patients in Arm C who are able to receive all treatment cycles before maintenance | Up to interim maintenance 2
  The feasibility of treating KMT2A-G patients with a high-risk ALL backbone and two cycles of blinatumomab (Arm C) will be assessed. Arm C treatment will be considered feasible for KMT2A-G patients if the proportion of KMT2A-G patients in Arm C who are able to receive all treatment cycles before maintenance (i.e., up to interim maintenance 2) is more than 76.8%. The proportion of patients receiving all cycles before Maintenance will be compared to 76.8% with a one-sample exact test of proportion with Type I error of 0.15.
3-year EFS of infants with KMT2A-G ALL treated on Arm C | From date of enrollment to treatment failure, first documented relapse following achievement of remission-1, occurrence of a second or secondary malignant neoplasm, or death, assessed up to 3 years
  The 3-year EFS rate from date of enrollment of KMT2A-G patients in Arm C will be estimated with the Kaplan-Meier method.
Pharmacokinetics (PK) of venetoclax in infants | On days 7, 10, and 14 of induction
  PK samples will be collected from patients enrolled in the safety phase of the study as well as from patients randomized to Arm B in the expansion phase who consent to participate, to determine the major secondary objective of characterizing the PK of venetoclax in infants. PK samples will be evaluated in batches and standard nonlinear mixed effect modeling will be used for model building and refinement of time-concentration data. After model refinement, a non-parametric bootstrap analysis will be performed reporting the 95% confidence intervals for each PK parameter.

OTHER OUTCOMES:
3-year EFS of infants with KMT2A-R ALL treated on Arm B | From date of randomization to treatment failure, first documented relapse following achievement of remission-1, occurrence of a second or secondary malignant neoplasm, or death, assessed up to 3 years
  Arm B, the 3-year EFS rate from date of randomization will be estimated, and will be compared to Arm A as described in the secondary objective, and to historical 3-year EFS. Comparison to historical rate will be based on a one-sample test of proportion with one-sided Type I error of 0.15.
Use of high-throughput sequencing (HTS) for MRD detection in infant ALL compared to centralized flow cytometry | Up to 3 years
  Pre-treatment HTS clonality and HTS MRD tracking results will be collected and compared to the required centralized flow cytometry-based MRD data to evaluate the feasibility and prognostic utility of HTS MRD evaluation in the infant ALL population.
PK of calaspargase pegol in infants with ALL | At completion of the trial, up to 3 years
  PK of calaspargase pegol will be analyzed by monitoring asparaginase activity levels. Once a PK model is developed for calaspargase pegol, standard regression analysis will be used to describe the relationship between drug exposure and asparaginase activity. Additionally, asparaginase-associated toxicities will be described for the entire study population and correlated with activity levels when possible. The result of this analysis will be an estimation of potential optimal exposure expected to yield the maximum efficacy while limiting toxicity. These analyses will be exploratory and descriptive.
Incidence of CD19-negative relapse and myeloid switch relapse with protocol therapy | At the time of relapse, up to 3 years
  For patients who experience relapse, will collect information regarding the immunophenotype of the leukemic blasts at time of relapse. Will report on the rate of CD19 negative relapse as well as myeloid switch relapse for all patients enrolled on study. This analysis will be exploratory and descriptive.
Impact of venetoclax in combination with chemotherapy on T-cell subsets and function | Prior to and following the first course of venetoclax
  BCL-2 inhibition is reported to alter T-cell subsets, including increased activation, enhanced cytotoxicity against leukemia cells and heightened resistance to cell death. Peripheral blood and bone marrow samples will be collected prior to and following the first course of venetoclax to evaluate effects on T-cell subsets and function following venetoclax exposure.
Feasibility of T-cell collection and success of T-cell manufacturing for infants with KMT2A-R ALL who receive chimeric antigen receptor (CAR) T-cell therapy | After coming off protocol therapy
  For patients that undergo T-cell collection, will collect data regarding the feasibility of T-cell collection in the context of protocol therapy. Additionally, for patients who proceed with CAR T-cell therapy after coming off protocol therapy, will collect data regarding the success of T-cell manufacturing, infusion and response to therapy in this young population, as the success of this subsequent therapy may be heavily impacted by the effect of protocol therapy on T-cell function. These analyses will be exploratory and descriptive.
Predictors of response and resistance to venetoclax and overall protocol therapy | Before and after venetoclax exposure, up to 3 years
  Will study the inter- and intra- patient variability in the expression of apoptotic proteins (e.g., BCL-2, MCL-1, BCL-XL) and apoptotic priming at diagnosis and identify changes that occur during induction therapy in relationship to venetoclax exposure. Will then determine whether the state of BCL-2 specific apoptotic priming correlates with outcome. Will also integrate genomic and molecular features (such as developmental state, signaling, epigenomic, transcriptomic, proteomic and metabolomic states) before and after venetoclax exposure, for those assays where this type of analysis is feasible, to determine biomarkers of response and resistance to therapy for infants with ALL.
Impact of subsequent anti-cancer therapy on overall survival | After coming off protocol therapy
  For all patients who remain in study follow-up after coming off protocol therapy, data will be collected regarding subsequent cancer directed therapies received as well as relapse and survival status in order to evaluate the impact of subsequent cancer directed therapy on the overall survival of patients enrolled on this study. These analyses will be exploratory and descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Erin H Breese, Principal Investigator — Children's Oncology Group
Locations (99):
- United States (98):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm